CLINICAL TRIAL: NCT06245668
Title: The Comparison of SaCoVLM™ Video Laryngeal Mask and LMA Supreme in Terms of Oropharyngeal Leak Pressure
Brief Title: SaCoVLM™ Video Laryngeal Mask Versus LMA Supreme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Assoc. Prof. Dr, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VLMSM5455
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia; Airway
Keywords: Supraglottic airway device

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer ('Urbaniak and Plous 2013')'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" ('Urbaniak and Plous 2013') tool to give each participation number to a random group with a 1:1 ratio.
  A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist who will administer the methods which group the patient is in immediately before administration. Researchers, patients, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SaCoVLM™ video laryngeal mask (Active Comparator): SaCoVLM™ video laryngeal mask
  Interventions: Device: SaCoVLM™ video laryngeal mask
- LMA Supreme (Active Comparator): LMA Supreme
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: SaCoVLM™ video laryngeal mask — The SaCoVLM™ video laryngeal mask will be placed directly into the hypopharyngeal space until resistance is felt, following the recommended instructions for use.
  Arms: SaCoVLM™ video laryngeal mask
Device: LMA Supreme — The LMA Supreme will be inserted directly by hand and placed into the hypopharyngeal space until resistance is felt, as per the recommended instructions for use.
  Arms: LMA Supreme

SUMMARY:
Our study aimed to compare two different laryngeal masks, SaCoVLM™ Video Laryngeal Mask and blind placement with LMA Supreme, in adult patients undergoing short elective surgeries. The aim is to optimize the use of commonly used laryngeal masks in clinical practice and examine the differences in oropharyngeal leak pressures.

DETAILED DESCRIPTION:
Laryngeal masks are alternative airway devices commonly used in anesthesia, serving both spontaneously breathing and ventilated patients. LMA Supreme, a second-generation laryngeal mask, has been widely used in routine anesthesia practices and short-duration procedures in our clinic. The advantage of second-generation masks is the presence of gastric access pathways, allowing for additional decompression of the stomach. SaCoVLM™ Video Laryngeal Mask also features a gastric access pathway. Placement of laryngeal masks requires attention to the anatomical features of the airway. Unsuccessful placement of a laryngeal mask can lead to issues such as throat pain, hoarseness, difficulty swallowing, airway obstruction, or leakage, as well as an increase in intragastric pressure due to gastric distention.

Our research is a prospective, randomized, controlled method study.The aim in this study is to reveal most accurate placement technique and device to transfer this method to clinical applications. Patients will be evaluated in two groups.

Group 1: Placement with SaCoVLM™ video laryngeal mask Group 2: Placement of the LMA Supreme with standard technique

After LMA Supreme and SaCoVLM™ video laryngeal mask placement, airway sealing pressures will be measured with appropriate technique. Airway tightness pressure measurement will be made with the technique accepted in the literature through the sensors in the anesthesia machine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* BMI < 35 kg/m2
* ASA (American Society of Anesthesiologists) physical score I/II
* Elective surgeries lasting less than 90 minutes

Exclusion Criteria:

* Patients who are expected to have a difficult airway
* Those with potential risk of regurgitation (severe reflux, presence of hiatal hernia)
* Those who will undergo head and neck surgery, laparoscopic surgery
* Those who will undergo surgery in the prone position
* Emergency surgical interventions
* Those requiring muscle relaxants
* Presence of oral abscess, pharyngeal pathology
* Those who have had an upper or lower respiratory tract infection in the last 4 weeks
* History of allergy to medications used
* Failure to obtain the consent of patients or their families

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | Immediately after the laryngeal mask is placed, before start of surgery
  Oropharyngeal leak pressure (OLP) will be measured by closing the adjustable pressure limiting valve on the anesthesia machine. The fresh gas flow was adjusted to 4 L/min. When the APL (Adjustable pressure limiting) valve was closed and manually ventilated. The leak sound that occurs during ventilation will be auscultated. The first peak airway pressure at which the leak occurs will be recorded as the oropharyngeal leak pressure.
  After successful insertion, laryngeal mask location will be evaluated with fiberoptic imaging.

SECONDARY OUTCOMES:
Assessment of Glottis Visualization Scores | Intraoperative period after the LMA insertion
  This will be assessed using five stages; Stage 1: Vocal cords not visible. Stage 2: Vocal cords and anterior epiglottis visible. Stage 3: Vocal cords and posterior epiglottis visible. Stage 4: Only vocal cords visible.
Peak Inspratuar Pressure and Plato Pressure | Intraoperative period
  Peak Inspratuar Pressure and Plato Pressure will be measured after the OLP measurement
Insertion time | Procedure (Time from LMA handling to first wave formation in capnography, assessed from the initiation of LMA handling until the detection of the first capnography wave.)
  Insertion time will be the time between picking up the device and successful placement
Number of attempts to place the device | Intraoperative period
  Number of attempts needed for successful placement will be recorded.
Blood pressure | Preoperatively, one minute after the induction, fifth minute and before removed laryngeal mask.
  Non-invasive blood pressure will measure blood pressure in millimeters of mercury.
Heart rate | Preoperatively, one minute after the induction, fifth minute and before removed laryngeal mask.
  Heart rate will be measured in beats per minute with an electrocardiography monitor.
Peripheral oxygen saturation | Preoperatively, one minute after the induction, fifth minute and before removed laryngeal mask.
  Peripheral oxygen saturation per minute will be measured by pulse oximetry
Complications | Intraoperative and postoperative day 1.
  The presence of complications that may be encountered after LMA removal will be investigated (Cough, Bucking, Laryngospasm, Aspiration, Desaturation(SpO2%< 90%), Need airway assist device(Nasal or oral airway), Blood on the surface of the cuff, hoarseness,sore throat)

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Dost, Assoc. Prof., Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Oba S, Turk HS, Isil CT, Erdogan H, Sayin P, Dokucu AI. Comparison of the Supreme and ProSeal laryngeal mask airways in infants: a prospective randomised clinical study. BMC Anesthesiol. 2017 Sep 5;17(1):125. doi: 10.1186/s12871-017-0418-z. PMID 28870163
- [Background] Van Zundert AAJ, Gatt SP, Kumar CM, Van Zundert TCRV, Pandit JJ. 'Failed supraglottic airway': an algorithm for suboptimally placed supraglottic airway devices based on videolaryngoscopy. Br J Anaesth. 2017 May 1;118(5):645-649. doi: 10.1093/bja/aex093. No abstract available. PMID 28510747
- [Background] Yan CL, Zhang YQ, Chen Y, Qv ZY, Zuo MZ. Comparison of SaCoVLM video laryngeal mask-guided intubation and i-gel combined with flexible bronchoscopy-guided intubation in airway management during general anesthesia: a non-inferiority study. BMC Anesthesiol. 2022 Sep 22;22(1):302. doi: 10.1186/s12871-022-01843-x. PMID 36138363
- [Background] Belena JM, Nunez M, Anta D, Carnero M, Gracia JL, Ayala JL, Alvarez R, Yuste J. Comparison of Laryngeal Mask Airway Supreme and Laryngeal Mask Airway Proseal with respect to oropharyngeal leak pressure during laparoscopic cholecystectomy: a randomised controlled trial. Eur J Anaesthesiol. 2013 Mar;30(3):119-23. doi: 10.1097/EJA.0b013e32835aba6a. PMID 23318811
- [Background] Yan CL, Zhang YQ, Chen Y, Qv ZY, Zuo MZ. To compare the influence of blind insertion and up-down optimized glottic exposure manoeuvre on oropharyngeal leak pressure using SaCoVLM video laryngeal mask among patients undergoing general anesthesia. J Clin Monit Comput. 2023 Apr;37(2):593-598. doi: 10.1007/s10877-022-00930-1. Epub 2022 Oct 29. PMID 36308611